CLINICAL TRIAL: NCT07151235
Title: A Controlled Human Environmental Study Evaluating the Impacts of Cognitive Functions During the Exposure of Simulated Wildfire-Related Air Pollution (WRAP).
Brief Title: Wildfire Related Air Pollution Exposure and Cognitive Function Pilot Study
Acronym: WRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jose Guillermo CEDENO LAURENT, ScD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro2025001070
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: wildfires; air pollution; ultrafine particles; cognitive function
MeSH Terms: conditions — Pemphigus and fogo selvagem

STUDY DESIGN:
Intervention Model Description: Participants will be exposed to two conditions (clean air and wildfire smoke) in random order.
Who Masked: Participant, Outcomes Assessor
Masking Description: outside laboratories processing blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure to simulated wildfire smoke, then exposure to clean air (Experimental): At the first study visit the subject undergoes a 1-hour chamber exposure to simulated wildfire smoke (300 ug/m3 Particulate Matter). After a 1-week washout period, the subject undergoes a 1-hour chamber exposure to clean air (0 ug/m3 PM).
  Interventions: Other: Simulated wildfire smoke exposure; Other: Clean Air exposure
- Exposure to clean air, then exposure to simulated wildfire smoke (Experimental): At the first study visit the subject undergoes a 1-hour chamber exposure to clean air (0 ug/m3 PM). After a 1-week washout period, the subject undergoes a 1-hour chamber exposure to simulated wildfire smoke (300 ug/m3 PM).
  Interventions: Other: Simulated wildfire smoke exposure; Other: Clean Air exposure

INTERVENTIONS:
Other: Simulated wildfire smoke exposure — 1 hour exposure to simulated wildfire smoke (300 ug/m3 PM)
Other: Clean Air exposure — 1 hour exposure to clean (HEPA-filtered) air (0 ug/m3 PM)

SUMMARY:
This study will examine how breathing wildfire-related air pollution (WRAP) for one hour affects healthy adults. The main question the study will answer if the effect of WRAP exposure on p-tau, a blood marker of cognitive decline. The changes in p-tau concentrations after exposure to WRAP will be compared to the changes in p-tau after exposure to clean air.

Participants will:

* Have 2 study visits - one visit with exposure to clean air and one visit with exposure to simulated wildfire smoke
* Have blood drawn before and after each exposure
* Complete cognitive tests and memory tasks before and after each exposure

DETAILED DESCRIPTION:
* Exposures will take place in a booth-like exposure chamber (1 x 0.7 x 1.8 m) with glass upper panels. One person will be exposed at a time.
* Simulated wildfire smoke will be generated by burning pine wood at a temperature that mimics smoldering combustion. The levels of smoke introduced into the exposure chamber are similar to those found during outdoor bonfires and wildfire events. The levels of particulate matter (PM) will be closely monitored during the exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non smoker
* Weight at least 110 pounds
* Between ages 18 and 40 years old

Exclusion Criteria:

* Claustrophobia or not comfortable in enclosed spaces.
* Colorblindness.
* Inability to hear verbal instructions.
* Cardiovascular disease which, in the opinion of the investigator, would elevate the participant's risk of adverse effects to WRAP exposure. This includes a history of stroke.
* Diabetes requiring the use of insulin.
* Pregnancy (A pregnancy test will be provided to you).
* Current asthma (an asthma attack within the past five years).
* History of childhood asthma.
* Medications which may affect cognition such as beta-blockers and CNS depressants.
* Respiratory symptoms in the previous 4 weeks (cough, wheezing, shortness of breath, etc.) which, in the opinion of the investigator, would elevate the participant's risk of adverse effects to WRAP exposure.
* Use of sedating cold/allergy medications in the previous week.
* Use of marijuana in the previous week.
* Consumption of alcohol in the previous 24 hours.
* Kidney or liver disease.
* Thyroid disease.
* High blood pressure.
* Cancer.
* Parkinson's disease.
* Pacemaker.
* Hay fever.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-09-18 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Changes in plasma P-tau 217 concentration from pre-exposure to post-exposure | Immediately before, immediately after each exposure
  Using blood samples collected pre- and post-exposure, the primary outcome will be assessed by measurement of plasma phosphorylated tau at threonine 217 (p-tau217) using an ultrasensitive immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Cedeno-Laurent, ScD, Principal Investigator — Rutgers, The State University of New Jersey: New Brunswick/Piscataway Campus
Locations (1):
- Rutgers-EOHSI, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2025-09-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT07151235/ICF_000.pdf